CLINICAL TRIAL: NCT06056934
Title: Retrospective Study of Protocol-based Pain Management in Elderly Patients With or Without Cognitive Frailty Hospitalized at UPOG for Fracture of the Upper Extremity of the Femur in 2022
Brief Title: Pain Management in Elderly Patients With or Without Cognitive Frailty Hospitalized "ALGOGER"
Acronym: ALGOGER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2023
Record Dates: First submitted 2023-06-22; First posted 2023-09-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Deterioration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, the standard treatment is to operate on patients suffering from a fracture of the upper end of the femur. The aim of treatment is to enable immediate mobilization and weight-bearing, and as rapid a return as possible to normal living conditions.

Surgery is the best treatment option. It maximizes the chances of functional recovery and, by stabilizing the fracture, reduces pain: it is the most effective and longest-lasting analgesic.

Adequate analgesia in elderly patients with femoral neck fractures has a beneficial effect. In particular, a lower probability of death has been shown in cervical fracture patients receiving opioids than those not receiving them.

Pain management is a matter of protocol in the UPOG department of the CHU de Nîmes.

Pain prevention appears to improve morbidity and mortality. Cognitive fragility, such as neurocognitive disorders, confusion or long-term use of psychotropic drugs, appear to be confounding factors in pain management.

The investigators therefore wished to observe whether the presence of cognitive fragility has an impact on pain management on the ward, despite protocol-based management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 75 years
* Hospitalized for a fracture of the upper extremity of the femur at the UPOG of the CHU de Nîmes during 2022

Exclusion Criteria:

* Opioid allergy
* No surgical management of fracture
* Long-term treatment with high-dose opiates
* Patient has objected to the use of his or her data.

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients hospitalized at UPOG for fracture of the upper end of the femur between January 1 and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Morphine sulfate equivalent rate in each group, mg/day | Pre-operative
  mg/day
Morphine sulfate equivalent rate in each group, mg/day | Early post-operative between Day 0 and Day 3
  mg/day
Morphine sulfate equivalent rate in each group, mg/day | Late post-operative between Day 4 and day 7
  mg/day

CONTACTS AND LOCATIONS:
Locations (1):
- GAULTIER, Nîmes, CHU de Nîmes, France